CLINICAL TRIAL: NCT07111429
Title: Evaluation of a Modified Clavien-Dindo Classification (COCG) of Stoma Complication in Cancer Patients: a Prospective, Registry-based, Non-randomized Trial (COCG-01 Trial) on Behalf of Chinese Ostomy Collaboration Group
Brief Title: Chinese Ostomy Collaboration Group (COCG) Clinical Study -SITI Classification
Acronym: COCG-SITI
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other); Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking Union Medical College Hospital (Other); Beijing New Journey Cancer Hospital (Unknown); Beijing Nanjiao Tumor Hospital (Unknown); Xuanwu Hospital, Beijing (Other); Beijing Hospital (Other Government); Hebei medical college fourth hospital (Unknown); China-Japan Union Hospital, Jilin University (Other); Jiangsu Province people hospital (Unknown); Jinzhou Medical University (Other); Shanxi Province Cancer Hospital (Other); Ruijin Hospital (Other); Changhai Hospital (Other); The Second Affiliated Hospital of Suzhou Medical University (Unknown); Tianjin People's Hospital (Other); Yantai Yuhuangding Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Zhejiang cancer University (Unknown); China-Japan Friendship Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Affiliated Drum Tower Hospital, Nanjing University (Unknown)
Responsible Party: Principal Investigator, Xiaokang Lei, Professor of Surgery, Chief physician, MD, Peking University Cancer Hospital & Institute
Other Study IDs: PekingUCHI
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Complication,Postoperative; Stoma
Keywords: stoma complications; SITI-CD Classification
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SITI-CD Classification of Stoma-related Complication in cancer patients: SITI-CD Classification of Stoma-related Complication in cancer patients
  Interventions: Diagnostic Test: Novel severity grading system of stoma-related complication in cancer patients

INTERVENTIONS:
Diagnostic Test: Novel severity grading system of stoma-related complication in cancer patients — Over 5000 stoma patients treated at 26 centers between 2022 and 2023 were classified according to SITI-CD Classification.

SUMMARY:
Colorectal cancer is an important cancer worldwide, and its incidence is increasing year by year. A large proportion of patients may require diverting stoma or even permanent stoma after surgery. Some of these patients will have a variety of stoma-related complications, which seriously affect the quality of life of patients. At present, the mainstream postoperative complication classification is the traditional CD classification, which is suitable for the classification of most postoperative complications. However, due to the unique anatomical characteristics of patients with stoma, the current CD classification system may not be suitable for the classification of patients with stoma-related complications. Therefore, we plan to establish a registry database of colorectal cancer patients with stoma, explore the attribution and incidence of stoma-related complications, and propose a new improved classification system, the SITI classification, on the existing CD classification, for verification and promotion.

DETAILED DESCRIPTION:
The complications related to stoma can be divided into five categories: skin complications near stoma (SKIN), abdominal incision complications at stoma (INCISION), abdominal wall fascia tunnel complications (abdominal Fascia/Muscular Tunnel complications), intestinal and mesenteric complications（Intestine）, and functional complications of ileostomy (Dehydration after IL). According to the actual situation of colostomy patients, the SITI classification is proposed to classify the complications from Grade Ia to V. The specific classification is as follows: Grade Ia, only need to observe, no treatment. Grade Ib, non-invasive treatment is required, and no drug is used. Grade IIa, invasive treatment without anesthesia, such as filling or local medication. Grade IIb, except for Grade IIa treatment, drugs, antibiotics, blood transfusion, etc. are used throughout the body. Grage IIIa, requiring intervention under local anesthesia. Grade IIIb, requiring intervention treatment of general anesthesia. Grade IVa, life threatening complications, including dialysis and single organ dysfunction. Grade IVb, complication of multiple organ dysfunction. Grade V, patient died. Classification, classification and grading can help ostomy therapists effectively identify and manage ostomy complications. The establishment of the database is convenient for researchers to explore the attribution of complications and the incidence of various types of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stoma after colorectal cancer resection.

Exclusion Criteria:

* Patients who don't want to be studied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colostomy after bowel cancer surgery were followed up for one year to understand the type and occurrence time of the complications of colostomy. Patients who were unwilling to accept the study were excluded
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of stoma complications in different SITI grades | 1year
  To understand the complications of different SITI grades, to clarify the rationality and feasibility of SITI grades, and to provide reasonable treatment for patients.

SECONDARY OUTCOMES:
Current status of surgeons' cognition of stoma complications | 2022-08 till 2023-08
  To understand the current situation of stoma complications in cancer patients, and to standardize the cognition of stoma classification among surgeons.It includes the classification criteria and treatment methods of stoma.
Global applicability of the SITI grades criteria | 2022-08 till 2023-08

CONTACTS AND LOCATIONS:
Overall Officials: LIN WANG, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Based on SITI classification, we will decide whether to conduct multicenter study or not